CLINICAL TRIAL: NCT00669448
Title: A Pilot Trial on the Effect of Mindfulness-based Cognitive Therapy Versus "Treatment as Usual" for Individuals With Multiple Chemical Sensitivities
Brief Title: A Pilot Trial on Effect of Mindfulness-based Cognitive Therapy for Individuals With Multiple Chemical Sensitivities (MCS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: The Danish Research Centre for Chemical Sensitivities, University Hospital, Gentofte
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID H-C-2007-0088; H-C-2007-0088
Record Dates: First submitted 2008-04-28; First posted 2008-04-30 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2008-04

CONDITIONS: Multiple Chemical Sensitivities
Keywords: Multiple chemical sensitivities; MCS; Mindfulness-based cognitive therapy; MBCT; Behavioural intervention; Stress; Illness perceptions; Pilot trial
MeSH Terms: conditions — Multiple Chemical Sensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Minfulness-based cognitive therapy — Mindfulness Based Cognitive Therapy (MBCT) is a group intervention that integrates elements from primarily Mindfulness-based Stress Reduction programme (MBSR)and cognitive therapy.The MBCT programme includes 2½ hours of training once a week for 8 weeks. In addition participants are encouraged to practice at home for up to 45 min per day, 6 days a week during the entire course.

SUMMARY:
OBJECTIVES

The objective is to evaluate the effect of an 8-week mindfulness-based cognitive therapy (MBCT) programme on psychological - and somatic symptoms, and illness perceptions in individuals with self- reported multiple chemical sensitivities.

PARTICIPANTS

Participants will be recruited among respondents to a survey on the consequences of self-reported symptoms related to inhalation of airborne chemicals conducted by the Danish Research Centre for Chemical Sensitivities.

DESIGN

The pilot trial is designed as a randomized trial on the effect of MBCT versus treatment as usual.

INTERVENTION

The MBCT programme includes 2½ hours of group training at the Psychiatric Centre, Rigshospitalet once a week for 8 weeks. Furthermore participants are encouraged to practice at home for up to 45 min per day, 6 days a week during the entire course.

OUTCOME MEASURES

Effect of MBCT will be estimated from individual scores on psychometric scales

DETAILED DESCRIPTION:
BACKGROUND

Multiple chemical sensitivities is a collective term used to describe illness from exposure to common environ-mental agents. A recent Danish population-based cross sectional study reported that 27% of the respondents reported various symptoms from exposure to common environmental agents. In 19% of the respondents symptoms had led to behavioral changes and in 3.3% of the respondents to adjustments in either social life or occupational conditions, and in 0.5% to adjustments in both social life and occupational conditions. Multiple chemical sensitivities is not acknowledged as a clinical diagnose in Denmark and the Danish Healthcare System has no clinical guidelines for management of people who report this type of illness.

OBJECTIVES

To evaluate the effect of an 8-week mindfulness-based cognitive therapy (MBCT) programme on psychological - and somatic symptoms, and illness perceptions in individuals with self- reported multiple chemical sensitivities.

PARTICIPANTS

Participants will be recruited among respondents to a survey on the consequences of self-reported symptoms related to inhalation of airborne chemicals conducted by the Danish Research Centre for Chemical Sensitives.

DESIGN

The pilot trial is designed as a randomized trial on the effect of MBCT versus treatment as usual. Eligible participants (n= 42) stratified by occupational status (e.g. employed/not employed) will be randomized to either intervention (MBCT) or treatment as usual.

INTERVENTION

The MBCT programme includes 2½ hours of group training at the Psychiatric Centre, Rigshospitalet once a week for 8 weeks. Furthermore participants are encouraged to practice at home for up to 45 min per day, 6 days a week during the entire course.

OUTCOME MEASURES

Effect of MBCT will be estimated from individual scores on the following psychometric scales: Symptom-Check List-92, The Brief Illness Perception Questionnaire, Perceived Stress Scale-10 and The Subjective Health Complaints-inventory. Estimations will be carried out at baseline, four weeks after start of MBCT programme, eight weeks after start of MBCT programme, and three months after ending the MBCT programme.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years,
2. Currently living in Zealand,
3. Self - reported adjustments of social life and/or occupational conditions due to symptoms related to inhalation of airborne chemicals,
4. Registered at the Danish Research Centre for Chemical Sensitivities because of self-reported symptoms attributed to common chemical scents,
5. Consulted the Al-lergy Clinic,
6. Rigshospitalet between 1990 and 2006 because of self-reported symptoms related to exposures to common environmental agents,
7. Informed consent

Exclusion Criteria:

1. Severe depression
2. Psychotic disorders
3. Medical treatment with antianxiety agents and antidepressants
4. Alcohol - or drug abuse
5. Previous participation in a MBCT programme
6. Lack of informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-04; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Symptom Checklist- 92 (SCL-92) | Baseline, four - and eight weeks after start of MBCT course, 3 months after ending MBCT course

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS-10) | Baseline, four - and eight weeks after start of MBCT course, three months after ending MBCT course
The subjective health complaints (SHC) inventory | Baseline, four- and eight weeks after start of MBCT course, 3 months after ending MBCT course
The Brief Illness Perception Questionnaire (Brief IPQ) | Baseline, four - and eight weeks after start of MBCT course, three months after ending MBCT course

CONTACTS AND LOCATIONS:
Overall Officials: Sine Skovbjerg, cand.san, Principal Investigator — The Danish Research Centre for Chemical Sensitivities
Locations (1):
- The Danish Research Centre for Chemical Sensitivities, Gentofte Municipality, Denmark